CLINICAL TRIAL: NCT04081298
Title: Adaptation and Evaluation of an Online and eHealth Diet and Physical Activity Program to Improve Cardiometabolic Health in Rural Latino Adults "Mi Vida Saludable en el Valle"
Brief Title: eHealth Diet and Physical Activity Program for the Improvement of Health in Rural Latino Cancer Survivors
Acronym: MiVSEEV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rachel Ceballos, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1005660; NCI-2019-05372 (Registry Identifier: NCI / CTRP); P30CA015704 (NIH); 10270 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
Keywords: Cancer Survivor
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Exercise; Health Promotion; Communication Devices for People with Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (eHealth program) (Experimental): Patients attend 6 online nutrition and PA education classes, cooking sessions, and participate in physical activities over 120 minutes each. Patients also receive text messages, electronic newsletters and have access to an interactive nutrition website.
  Interventions: Behavioral: Health Education; Other: Physical Activity; Other: Health Promotion and Education: Text Messages; Other: Health Promotion and Education: Web Site; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Health Education — Attend nutrition and PA classes, and cooking sessions
Other: Physical Activity — Participate in physical activities
Other: Health Promotion and Education: Text Messages — Receive motivational text messages
  Other Names: Text
Other: Health Promotion and Education: Web Site — Given access to nutrition website
  Other Names: Internet Website; Website; www-website
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how to improve the diet quality and physical activity level of Latino cancer survivors living in rural areas. The recommendation to eat a high-quality diet and engage in moderate-to-vigorous physical exercise may reduce cancer risk, improve cancer survival rate, and reduce associated conditions. However, it is not well understood how best to teach cancer survivors, especially Latino cancer survivors living in rural areas, to achieve and maintain diet and physical activity. Understanding how to build a culturally appropriate education that is effective may improve the diet quality and physical activity level of Latino cancer survivors.

DETAILED DESCRIPTION:
OUTLINE:

Patients attend 6 online nutrition and physical activity (PA) education classes, cooking sessions, and participate in physical activities over 120 minutes each. Patients also receive text messages, electronic newsletters and have access to an interactive nutrition website.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-identify as being at least 18 years of age or older
* Participants must self-identify as Latino
* Participants must be a resident of the Lower Yakima Valley (LYV) and anticipate remaining in the LYV for at least 1 year
* Participants must speak Spanish or English and fully understand Spanish for online group sessions
* Participants must self-identify as having a medical history of hypertension
* Participants must self-identify as having a medical history of diabetes
* Participants must self-identify as having a medical history of cardiovascular disease
* Participants must self-identify as having a medical history of obesity, as defined by a body mass index (BMI) of > 30 kg/m^2
* Participants must self-identify as having a medical history of cancer (excluding non-melanoma skin cancer). All other cancer types will be included provided
* There is no evidence of recurrent or metastatic disease
* The patient has not received a bone marrow, stem cell, or cord blood transplant
* For cancer survivors, participants must self-identify as being at least 60 days post final chemotherapy, biologic therapy, or radiation therapy treatment and/or surgery. Current use of hormonal therapy is permitted (e.g., tamoxifen and aromatase inhibitors)
* Participants must be willing and able to receive text messages via cellphone for 3-6 months
* Participants must be willing and able to attend six 120-minute online group sessions
* Participants must be willing to complete the surveys, and diet/PA assessments
* Participants who report having been told by a health professional they have diabetes or cardiovascular disease must provide a clearance from their physician for participation
* Participants must consume < 5 servings of fruits and vegetables per day and/or engage in < 150 minutes per week of moderate to vigorous physical activity, as assessed by brief questionnaires
* Participants must have an Eastern Cooperative Oncology Group (ECOG) scale of performance status score of 0 or 1 for performance status. These scales and criteria are commonly used by doctors and trained research staff to assess a person's daily living abilities. These scales and criteria are commonly used by doctors and trained research staff to assess a person's daily living abilities. Scores of 0 and 1 corresponds to being fully active, able to carry on all pre-disease performance without restriction; and restricted in physically strenuous activity but ambulatory and able to carry our work of a light or sedentary nature, respectively
* Ability to understand and the willingness to sign an online informed consent document * Depending on preference, the consent will be provided in English or Spanish

Exclusion Criteria:

* Participants must not be active smokers within the past 30 days. Active smoking is defined as any smoking, even a puff. Participants who smoke are much less likely to engage in healthy lifestyle behaviors, and it is probably more important for participants to stop smoking than it is to change their dietary patterns. If identified as a smoker, the individual will be referred the Centers for Disease Control and Prevention (CDC) "Quit Now" phone line which supports smoking cessation, or the National Institutes of Health (NIH) quit support website SmokeFree.gov which are both available in English and Spanish
* Women must not be pregnant at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Ceballos, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was paused April 2020 due to the pandemic. Because we had not reached the number needed to begin our first intervention cohort and pandemic protocols halted our in-person study design, the project was paused. We revised the study design and began recruitment again with a new online version of the protocol, recruitment protocols, and participant eligibility on 9/16/2021. The revised protocol concluded on 2/25/2022.
Pre-assignment Details: As this was a single arm study, participants were not assigned to any arm or group.
Groups:
- eHealth Diet and Physical Activity Education and Communication: This is a single arm feasibility study to assess a culturally tailored eHealth diet and physical activity education and communication program for rural Latino adults with a history of hypertension, diabetes, cardiovascular disease, cancer, and/or obesity in the Lower Yakima Valley in Washington State.
Period: Overall Study
Arm/Group | eHealth Diet and Physical Activity Education and Communication
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: This is a single arm feasibility study to assess a culturally tailored eHealth diet and physical activity program for rural Latino adults with a history of hypertension, diabetes, cardiovascular disease, cancer, and/or obesity in the Lower Yakima Valley.
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Other | 7
  Race: White | 12
  Race: Black or African American | 1
Region of Enrollment [Count of Participants; unit: Participants] — Because this is a feasibility study, retention was measured. The overall number of baseline participants was 20 and 19 were included in the final analyses. This is due to a loss to follow up of 1 participant and reflects a 95% retention rate.
  Participants
    United States | 20
Place of Birth [Count of Participants; unit: Participants] — Indicates if participant is born in the U.S. vs foreign-born
  Participants
    U.S born | 12
    Foreign born | 8
Years of education [Mean (Standard Deviation); unit: years] | 12.3 (3.8)
Body Mass Index [Mean (Standard Deviation); unit: kg/m-squared] | 33.6 (7.2)
Married or Living With Partner [Count of Participants; unit: Participants]
  Married or Living with Partner | 10
  Living Alone | 10
Number of Household Members [Mean (Standard Deviation); unit: Household Members] | 3.9 (2.1)
Use of Electronic Benefit Transfer/Supplemental Nutrition Assistance Program [Count of Participants; unit: Participants] | 3
Employment Status [Count of Participants; unit: Participants]
  Employed (FT or PT) | 11
  Unemployed | 9
Languages Spoken at Home [Count of Participants; unit: Participants]
  Only Spanish | 6
  More Spanish than English | 2
  Both Spanish and English Equally | 4
  More English than Spanish | 8
Clinical Diagnosis [Count of Participants; unit: Participants]
  Diabetes | 8
  Hypertension | 6
  Cholesterol | 3
  Liver Disease | 2
  Gastrointestinal Problems | 3
  Cancer | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Retention
Description: Number of participants that completed the follow-up (3 month) data collection. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3-months
Measure: Count of Participants; unit: Participants
Groups:
- Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication: Patients attend 6 online nutrition and PA education classes, cooking sessions, and participate in physical activities over 120 minutes each. Patients also receive text messages, electronic newsletters and have access to an interactive nutrition website.
  Health Education: Attend nutrition and PA classes, and cooking sessions
  Physical Activity: Participate in physical activities
  Health Promotion and Education: Text Messages: Receive motivational text messages
  Health Promotion and Education: Web Site: Given access to nutrition website
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants | 19

2. Primary Outcome: Feasibility: Adherence for Text Messages
Description: Number of participants who responded to 1 or more text messages. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 20
Participants | 10

3. Primary Outcome: Feasibility: Adherence of Grocery Deliveries
Description: Number of times participant received all 6 grocery deliveries. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 20
Participants | 19

4. Primary Outcome: Feasibility: Adherence for Online Sessions
Description: For the purpose of this feasibility study, participants who completed at least 3 of the 6 online sessions were assessed. Participants attend 6 online nutrition and PA education classes, cooking sessions, and participate in physical activities over 120 minutes each. Patients also receive text messages, electronic newsletters and have access to an interactive nutrition website Health Education: Attend nutrition and PA classes, and cooking sessions Physical Activity: Participate in physical activities This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants | 13

5. Primary Outcome: Feasibility: Acceptability of Cooking Sessions
Description: Acceptability of the cooking sessions was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  Cooking sessions were somewhat or very helpful | 18
  Cooking sessions were somewhat or not very helpful or not at all helpful | 1

6. Primary Outcome: Feasibility: Acceptability of Recipes
Description: Acceptability of recipes was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication: Patients attend 6 online nutrition and PA education classes, cooking sessions, and participate in physical activities over 120 minutes each. Patients also receive text messages, electronic newsletters and have access to an interactive nutrition website.
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  Recipes were somewhat or very helpful | 19
  Recipes were somewhat or not at all helpful | 0

7. Primary Outcome: Feasibility: Acceptability Nutrition and Physical Activity Sessions
Description: Acceptability of the nutrition and physical activity sessions was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  Nutrition and physical activity sessions were somewhat or very helpful | 19
  Nutrition and physical activity sessions were not very helpful or not at all helpful | 0

8. Primary Outcome: Feasibility: Acceptability of Nutrition Text Messages
Description: Acceptability of the nutrition text messages was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  nutrition text messages were somewhat or very helpful | 18
  nutrition text messages were not very helpful or not at all helpful | 1

9. Primary Outcome: Feasibility: Acceptability of Physical Activity Text Messages
Description: Acceptability of physical activity text messages was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  physical activity text messages were somewhat or very helpful | 18
  physical activity text messages were not very helpful or not at all helpful | 1

10. Primary Outcome: Feasibility: Acceptability of Website
Description: Acceptability of the website was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery.This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  Website was somewhat or very helpful | 12
  Website was not very helpful or not at all helpful | 7

11. Primary Outcome: Feasibility: Acceptability of FITBit
Description: Acceptability of the FITBit was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery.This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  Fitbits were somewhat or very helpful | 16
  Fitbits were not very helpful or not at all helpful | 3

12. Primary Outcome: Feasibility: Acceptability of Monthly check-in Calls
Description: Acceptability of monthly check-in calls was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  Monthly checking in calls were somewhat or very helpful | 18
  Monthly checking in calls were not very helpful or not at all helpful | 1

13. Primary Outcome: Feasibility: Acceptability of Contact With Study Staff
Description: Acceptability of contact with study staff was assessed during the exit interview. The exit interview asked participants to respond to a series of 15-questions assessing the helpfulness of each intervention component (e.g., online session, FITBit, e-communications, etc). Response options include a 6-item Likert scale (1=not at all helpful to 5=very helpful). A space for written-qualitative responses was also provided to allow the participant to provide information about the context and recommendations related to the intervention components/delivery. This feasibility study has primary outcomes that are descriptive in nature and do not include statistical analyses. The outcome measure data table provide the feasibility results for the project.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
Participants
  Contact with study staff was somewhat or very helpful | 18
  Contact with study staff was not very helpful or not at all helpful | 1

14. Secondary Outcome: Nutrition Preferences: Fruit and Vegetables
Description: Nutrition preferences were measured using 17-questions adapted from a battery developed and validated by the study team. The battery is titled "The Preferences and Self-Efficacy of Diet and Physical Activity Behaviors Questionnaires for Latinas" (preparing manuscript for submission). Participants were asked to rate their like or dislike for 11 specific fruits or vegetables (e.g., green cabbage, kale, turkey or veggie burgers, foods made with oil instead of butter or lard). For each fruit or vegetable listed they were asked to rate on a 5 point likert scale with 1=strongly dislike to 5=strongly like or respond with "never tried it"=0. Scores are averaged across the 17 items. Higher scores are considered a better outcome.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
score on a scale
  Baseline | 3.80 (0.89)
  3 month follow-up | 4.04 (0.41)
Statistical Analysis 1: Comparison: Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication; Test type: Equivalence — feasibility assessment; p = 0.24, Paired sample t-test — The threshold for statistical significance is p=0.05. (feasibility assessment); Mean Difference (Final Values) = 0.24, Standard Deviation 0.80

15. Secondary Outcome: Nutrition Self-Efficacy
Description: Nutrition Self-efficacy was measured using 11-questions from a battery developed and validated by the study team. The battery is titled "The Preferences and Self-Efficacy of Diet and Physical Activity Behaviors Questionnaires for Latinas" (preparing manuscript for submission). Participants were asked to rate thow confident they are in their ability to engage in healthy dietary behaviors for one month. For each behavior listed they were asked to rate on a 5 point likert scale with 1=not at all confident to 5=extremely confident. Scores are averaged across the 11 items. Higher scores are considered a better outcome.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
score on a scale
  Baseline | 3.20 (0.76)
  3 month follow-up | 3.34 (0.69)
Statistical Analysis 1: Comparison: Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication; Test type: Equivalence — feasibility assessment; p = 0.43, paired t-test — The threshold for statistical significance was p=0.5 (feasibility assessment); Mean Difference (Final Values) = 0.14, Standard Deviation 0.78

16. Secondary Outcome: Nutrition Knowledge
Description: Nutrition knowledge was a single question. The value reflects a change in the percent of women who correctly answered the targeted number of daily serving intake of fruits and vegetables at baseline compared to 3-month follow-up. The correct answer was 5-9 servings per day.
Time Frame: Change in correct nutrition knowledge response from baseline to 3 month follow-up
Population: McNemar's test for binary measures.
Measure: Number; unit: change in % of correct responses
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
change in % of correct responses | 21
Statistical Analysis 1: Comparison: Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication; Single arm pre-post comparison at baseline and 3-month follow-up (feasibility study); Test type: Equivalence — McNemar's test evaluates equivalence between nominal groups. Power not calculated as this is a feasibility study with small sample size; p = 0.10, McNemar

17. Secondary Outcome: Physical Activity Preferences
Description: Physical Activity preferences were measured using 8-questions from a battery developed and validated by the study team. The battery is titled "The Preferences and Self-Efficacy of Diet and Physical Activity Behaviors Questionnaires for Latinas" (preparing manuscript for submission). Participants were asked to rate their like or dislike for 8 specific types of physical activity (e.g., doing housework with vigorous effort, dancing in a group setting, playing with children with vigorous effort). For each activity listed they were asked to rate on a 5 point likert scale with 1=strongly dislike to 5=strongly like or respond with "never tried it"=0. Scores are averaged across the 8 items. Higher scores are considered a better outcome.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
score on a scale
  Baseline | 3.47 (0.70)
  3 month follow-up | 3.66 (0.55)
Statistical Analysis 1: Comparison: Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication; Test type: Equivalence — feasibility assessment; p = 0.20, paired-sample t-test — The threshold for statistical significance was p=0.5 (feasibility assessment); Mean Difference (Final Values) = 0.20, Standard Deviation 0.65

18. Secondary Outcome: Physical Activity Self-Efficacy
Description: Physical Activity Self-Efficacy: Self-efficacy was measured using 5-questions from a battery developed and validated by the study team. The battery is titled "The Preferences and Self-Efficacy of Diet and Physical Activity Behaviors Questionnaires for Latinas" (preparing manuscript for submission). Participants were asked to rate how confident they are in their ability to engage in healthy physical activity behaviors given certain conditions (e.g., when you can't notice any improvements in your fitness, when you have many other demands on your time, when you feel a little stiff or sore) for one month. For each behavior listed they were asked to rate on a 5 point likert scale with 1=not at all confident to 5=extremely confident. Scores are averaged across the 5 items. Higher scores are considered a better outcome.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
score on a scale
  Baseline | 3.12 (0.69)
  3 month follow-up | 3.18 (0.64)
Statistical Analysis 1: Comparison: Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication; Test type: Equivalence — paired sample t-test (feasibility assessment); p = 0.71, paired sample t-test; Mean Difference (Final Values) = 0.06, Standard Deviation 0.73

19. Secondary Outcome: Self-Reported Physical Activity: Time Sitting
Description: Self-reported physical activity reflects change in time spent sitting (minutes/day). NOTE: The outcomes are reported as a change score (value at 3 months minus value at baseline)
Time Frame: Baseline and 3 month follow-up
Measure: Mean (Standard Deviation); unit: change in mean (minutes/day)
Arm/Group | Health Services Research (eHealth Program)
Number analyzed (Participants) | 19
change in mean (minutes/day) | -3.6 (128.7)
Statistical Analysis 1: Comparison: Health Services Research (eHealth Program); Single arm pre-post comparison at baseline and 3-month follow-up (feasibility study); Test type: Equivalence — The analysis is an equivalence analysis of change (H1) in mean value from baseline to 3 month follow-up. Power was not calculated for this analysis because this is a feasibility study. The sample size is not large enough to approach appropriate power; p = 0.94, paired-sample t-test

20. Secondary Outcome: Self-Reported Physical Activity: Walking
Description: Self-reported physical activity: walking (MET-minutes/week). NOTE: METs=metabolic equivalent of task. Walking in this case is defined as a light activity equivalent to < 3 METs. The outcomes are reported as a change score (value at 3 months minus value at baseline).
Time Frame: Baseline and 3 month-follow-up
Measure: Mean (Standard Deviation); unit: change in mean (MET-minutes/week)
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
change in mean (MET-minutes/week) | 490 (907)
Statistical Analysis 1: Comparison: Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication; Test type: Equivalence — The analysis is an equivalence analysis of change (H1) in mean value from baseline to 3 month follow-up using a paired-sample t-test. Power was not calculated for this analysis because this is a feasibility study. The sample size is not large enough to approach appropriate power; p = 0.03, paired-sample t-test

21. Secondary Outcome: Self-Reported Physical Activity: Moderate to Vigorous Physical Activity
Description: Self-reported physical activity includes moderate to vigorous physical activity (MET-minutes/week).
  NOTE: METs=metabolic equivalent of task. Moderate to Vigorous Physical Activity is considered activities estimated at 3 or more METs. The outcomes are reported as a change score (value at 3 months minus value at baseline)
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Deviation); unit: change in mean (MET-minutes/week)
Arm/Group | Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication
Number analyzed (Participants) | 19
change in mean (MET-minutes/week) | -1024 (4709)
Statistical Analysis 1: Comparison: Health Services: Single Arm Feasibility Online Diet and Physical Activity and eHealth Communication; Test type: Equivalence — [test comment as in outcome 20, analysis 1]; p = 0.36, paired-sample t-test

ADVERSE EVENTS:
Time Frame: 3 month intervention delivery period.
Description: No adverse events to report.
Groups:
- eHealth Diet and Physical Activity Program: This is a single arm feasibility study to assess a culturally tailored eHealth diet and physical activity education and communication program for rural Latino adults with a history of hypertension, diabetes, cardiovascular disease, cancer, and/or obesity in the Lower Yakima Valley in Washington State.
Arm/Group | eHealth Diet and Physical Activity Program
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04081298/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT04081298/ICF_000.pdf